CLINICAL TRIAL: NCT04124211
Title: Fecal Microbiome Transplantation (FMT) for Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Affiliated Hospital of Southern Medical University (Other Government)
Collaborators: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Jie Shen, MD, Director of Endocrinology, The Third Affiliated Hospital of Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYSY-NFM; 2018-lunshen-017 (Other: No.3 Affiliated Hospital of SMU)
Record Dates: First submitted 2019-08-23; First posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Type 1 Diabetes
Keywords: Fecal Microbiome Transplantation (FMT)
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT Arm (Experimental): 10 Participants will be enrolled in this arm to receive FMT treatment
  Interventions: Biological: Fecal Microbiota Transplantation (FMT)

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation (FMT) — FMT will be performed through transendoscopic enteral tubing (TET) within one week during treatment period

SUMMARY:
This study intends to reconstruct intestinal micro-ecology through fecal Microbiome transplantation (FMT) technology, to treat patients with type 1 diabetes, and combine intestinal Metagenomics and 16s rRNA sequencing technology to study the relevant mechanism of intestinal micro-ecology for the treatment of type 1 diabetes.

DETAILED DESCRIPTION:
Type 1 diabetes is an organ-specific autoimmune disease based on islet beta cell-specific destruction and absolute insulin deficiency. Studies on the pathogenesis of intestinal flora and type 1 diabetes have shown that as an "endocrine organ", intestinal microbes play an important role in regulating the secretion of the body. Bacteria in the intestine can not only directly synthesize hormones or hormone-like compounds, but also regulate the synthesis and secretion of corresponding hormones in the widely distributed intestinal endocrine cells, thereby participating in the regulation of various biological functions in the human body. This study uses fecal microbiome transplantation (FMT) to explore another potential treatment for type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* (1) Type 1 diabetes patients.
* (2) Age between 18 and 65 years old, regardless of gender.
* (3) No serious comorbidities.
* (4) Accept and suitable for endoscopic catheterization (TET) and fecal transplantation (FMT).
* (5) Can receive follow-up and follow-up examinations on time. (6) Subjects need to sign an informed consent form.

Exclusion Criteria:

* (1) Systematic application of glucocorticoids, other immunosuppressive drugs or biological immune modulators, antibiotics, probiotics, and other microecological agents to alter intestinal motility within 6 months prior to enrollment.
* (2) An infection that is active.
* (3) Combined with irritable bowel syndrome, inflammatory bowel disease, celiac disease, and other chronic gastrointestinal diseases, the condition has not been controlled.
* (4) Chronic diseases such as cerebrovascular disease, cardiovascular disease, and diabetic autonomic neuropathy.
* (5) Pregnancy or with a pregnancy plan
* (6) severe organ dysfunction (including decompensated cirrhosis, malignant tumors, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-08-25 (Actual); Primary Completion 2020-03-10 (Estimated); Study Completion 2020-03-10 (Estimated)

PRIMARY OUTCOMES:
Changes in mean amplitude of glycemic excursion (MAGE) | 24 Weeks
  Dates from Continuous glucose monitoring system
Changes in standard deviation of blood glucose (SDBG) | 24 Weeks
  Dates from Continuous glucose monitoring system
Changes in hemoglobin A1c (HbA1c) | 24 Weeks
  Dates from blood chemistry test
Safety of FMT | 24 Weeks
  Number of all participants with treatment-related adverse events as assessed by CTCAE v4.03

SECONDARY OUTCOMES:
Changes in 24h mean blood glucose(MBG) | 24 Weeks
  Dates from Continuous glucose monitoring system
Changes in percentage of time of blood glucose(PT) | 24 Weeks
  Dates from Continuous glucose monitoring system
Changes in mean absolute glucose(MAG) | 24 Weeks
  Dates from Continuous glucose monitoring system
Changes in standard deviation of blood glucose(SDBG) | 24 Weeks
  Dates from Continuous glucose monitoring system
Changes in coefficient of variation(CV) | 24 Weeks
  Dates from Continuous glucose monitoring system
Changes in high blood glucose index(HBGI) | 24 Weeks
  Dates from Continuous glucose monitoring system
Changes in low blood glucose index(LBGI) | 24 Weeks
  Dates from Continuous glucose monitoring system
Changes in effective blood glucose fluctuations in frequency(NGE) | 24 Weeks
  Dates from Continuous glucose monitoring system
Changes in glycated albumin (GA) | 24 Weeks
  Dates from blood chemistry test
Changes of serum C-peptide (fasting, 30min after meal, 120min after meal) | 24 Weeks
  Dates from blood chemistry test
Assessment of diabetes antibodies | 24 Weeks
  Assessment of diabetes antibodies including Islet Cell Cytoplasmic Autoantibodies (ICA), Insulin Autoantibodies (IAA), Glutamic Acid Decarboxylase Autoantibodies (GADA), Insulinoma-Associated-2 Autoantibodies (IA-2A), and Zinc Transporter-8 Autoantibodies (ZnT8A);
Changes in intestinal microbiome profile | 24 Weeks
  Changes in intestinal microbiome profile by 16s rRNA sequencing and metagenomics.
Changes in Peripheral Blood Stem Cell (PBMC) | 24 Weeks
  Dates from blood test
Changes in body weight to calculate body mass index (BMI) | 24 Weeks
  Dates from physical examination
Pathological changes of intestinal mucosa | 24 Weeks
  Changes in intestinal mucosa profile by enteroscopy
Changes in blood pressure | 24 Weeks
  Dates from physical examination
Changes in oral mucosal bacteria colonization | 24 Weeks
  Changes in oral mucosal bacteria by 16s rRNA sequencing and metagenomics.
Changes in urine microalbumin | 24 Weeks
  Dates from urine test
Blood chemistry panel | 24 Weeks
  Changes in the results of blood chemistry tests including complete blood count, diabetic autoantibodies, serum C peptide, insulin, blood glucose, routine urine, urinary microalbumin, routine stool, liver function, renal function, seven ions, myocardial enzymes, six glycolipids, glycated hemoglobin and glycosylated serum albumin before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Shen, MD, Principal Investigator — The Third Affiliated Hospital of Southern Medical University
Locations (1):
- The third affiliated hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No